CLINICAL TRIAL: NCT00005764
Title: Glaxo Wellcome Trial to Assess the Regression of Hyperlactatemia and to Evaluate the Regression of Established Lipodystrophy in HIV-1-Positive Subjects (TARHEEL)
Brief Title: A Study of Increased Lactic Acid and Abnormal Fat Distribution in HIV-Positive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 238T; ESS40010
Record Dates: First submitted 2000-05-30; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-06

CONDITIONS: HIV Infections; Lipodystrophy
Keywords: HIV-1; Zalcitabine; Didanosine; Drug Therapy, Combination; Zidovudine; Stavudine; Lamivudine; Blood; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Lipodystrophy; Combivir; Lactic Acid; abacavir
MeSH Terms: conditions — HIV Infections; Lipodystrophy | interventions — lamivudine, zidovudine drug combination; abacavir; Lamivudine

INTERVENTIONS:
Drug: Lamivudine/Zidovudine
Drug: Abacavir sulfate
Drug: Lamivudine

SUMMARY:
The purpose of this study is to see if the findings of increased lactic acid and abnormal fat distribution get better when d4T is replaced with abacavir, abacavir plus lamivudine, or Combivir (a pill containing lamivudine plus zidovudine) in HIV-positive patients taking anti-HIV therapy including stavudine (d4T).

DETAILED DESCRIPTION:
Patients are allocated as follows: a) zidovudine-naive patients switch Combivir for d4t and b) zidovudine-experienced or -intolerant patients switch abacavir for d4t. Providers may choose between Combivir or abacavir as a switch for d4t when screening lactate levels are 2.2 mmol/L or more. Additionally, providers may choose to switch a maximum of 2 drugs, one of which must be d4t, in the regimen. Each patient receives 48 weeks of therapy. Visits are made at Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, and 48. Tests, including biopsies, are performed to measure changes in body fat distribution and changes in lactate levels. Virologic and immunologic outcomes, changes in physical signs of lipodystrophy, changes in self-reports of health-related quality-of-life survey and the Body Image Questionnaire, changes in lipid profile and other markers of metabolism, and safety parameters are evaluated also.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Are at least 18 years old.
* Agree not to have intercourse 2 weeks before, during, and 2 weeks after study or agree to use effective methods of birth control.
* Have had HIV-1 RNA levels less than 400 copies/ml on the 2 most recent measurements.
* Have at least 1 of the following situations:
* (a) at least 1 of the following: (1) decrease in facial fat, (2) decrease in fat in lower limbs, or (3) decrease in fat in buttocks area; or
* (b) an increase in lactate level greater than 2.2 mmol/L at the screening visit plus at least 1 of the following: (1) decrease in facial fat, (2) decrease in fat in lower limbs, or (3) decrease in fat in the buttocks area; or
* (c) an increase in lactate level greater than 2.2 mmol/L at screening visit plus at least 2 of the following: (1) shortness of breath, (2) weakness, (3) fast heartbeat, (4) recent weight loss (10 lbs. within the past 2 months), (5) pain and/or bloating in the abdomen, (6) nausea and/or vomiting and/or lack of appetite; or
* (d) lactate level greater than 3.2 mmol/L at the screening visit.
* Are able to read at a sixth-grade level.
* Have taken d4T consistently for the 6 months before entering study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have diabetes or kidney failure.
* Have any condition that makes them unable to participate in this study.
* Are unable to take medications by mouth.
* Have serious medical conditions, such as congestive heart failure or other heart disease, which would affect the safety of the patient.
* Are taking or have taken abacavir plus Retrovir or Combivir.
* Are pregnant or breast-feeding.
* Are enrolled in other clinical studies.
* Have had a reaction to or are unable to take abacavir and have taken Retrovir in the past.
* Have taken hydroxyurea within the past 3 days or plan to take this drug during the study.
* Have had chemotherapy or radiation therapy within 4 weeks prior to screening visit (except for local treatment for Kaposi's sarcoma) or plan to have such treatment during the study.
* Have taken drugs that affect the immune system, such as systemic corticosteroids, interleukins, vaccines, or interferons, within 4 weeks prior to the screening visit.
* Have had an HIV vaccine within 3 months of the screening visit.
* Have taken recombinant Human Growth Hormone (r-hGH), megestrol acetate, medicines containing oxandrolone, oxymetholone, nandrolone, DHEA, or other testosterone derivatives, or glucocorticoids or other systemic steroids (except inhaled and topical steroids) in the last 4 months or plan to take these drugs during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2000-05

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - THE Clinic, Los Angeles, California
  - Tower Infectious Disease Med Ctr, Los Angeles, California
  - St Lukes Medical Group, San Diego, California
  - UCSD Treatment Ctr, San Diego, California
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - North Broward Hosp District / HIV Clinical Research, Fort Lauderdale, Florida
  - Duval County Health Department, Jacksonville, Florida
  - Infectious Disease Research Institute Inc, Tampa, Florida
  - Northstar Med Clinic, Chicago, Illinois
  - Jersey Shore Med Ctr, Neptune City, New Jersey
  - South Jersey Infectious Diseases Inc, Somers Point, New Jersey
  - Infectious Disease Specialists of NJ, Union, New Jersey
  - Infectious Diseases Assoc of Brooklyn, Brooklyn, New York
  - Long Island College Hospital, Brooklyn, New York
  - Mt Vernon Hospital, Mount Vernon, New York
  - Dr Lawrence Fontana, New York, New York
  - Liberty Medical / Cabrini Hospital / Dept of Infec Diseases, New York, New York
  - Howard Grossman, New York, New York
  - Boriken Neighborhood Health Center, New York, New York
  - Bronx Veterans Affairs Med Ctr, The Bronx, New York
  - Univ of North Carolina / SOCA, Chapel Hill, North Carolina
  - Summa Health System, Akron, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - Philadelphia Veterans Administration Med Ctr, Philadelphia, Pennsylvania
  - Anderson Clinical Research, Pittsburgh, Pennsylvania
  - Central Texas Clinical Research, Austin, Texas
  - Gathe, Joseph, M.D., Houston, Texas
  - Diversified Med Practices, PA, Houston, Texas
  - Univ of Texas / Med School at Houston, Houston, Texas
  - Hampton Roads Med Specialists, Hampton, Virginia
  - Swedish Med Ctr, Seattle, Washington